CLINICAL TRIAL: NCT06593392
Title: KOR-PED-202 An Open-label, Single-arm Study to Evaluate the Safety and Tolerability of Intravenous Difelikefalin in Adolescents Aged 12 to 17 Years on Haemodialysis With Moderate-to-Severe Pruritus
Brief Title: Safety and Tolerability of Difelikefalin in Adolescents on Haemodialysis With Moderate-to-Severe Pruritus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vifor Fresenius Medical Care Renal Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOR-PED-202
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Pruritus; Chronic Kidney Diseases
Keywords: Chronic kidney disease associated pruritus
MeSH Terms: conditions — Pruritus; Renal Insufficiency, Chronic | interventions — difelikefalin

STUDY DESIGN:
Intervention Model Description: Open label single arm phase IIb clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Difelikefalin

INTERVENTIONS:
Drug: Difelikefalin — The study includes a screening period of up to 4 weeks (including a 7-day run-in period during the week prior to enrolment), a study treatment period of 12 weeks, and a safety follow-up visit at 7 (up to 10) days after EoT. Total study duration for a single participant is up to 17 to 18 weeks.

SUMMARY:
Rationale:

* People with long term kidney disease who are on haemodialysis (a procedure for removing waste products from the blood) commonly develop a condition that makes their skin very itchy.
* Difelikefalin is a medicine that can treat the itching related to long term kidney disease.
* Clinical studies have shown difelikefalin to reduce itching in adults on haemodialysis, while being safe and tolerable.
* The current study is being done in adolescents aged 12 to 17 years on haemodialysis who have moderate to severe itching related to long term kidney disease to assess if difelikefalin is safe in this age group.

The aims of the study are:

Main aim: To assess the safety of difelikefalin in adolescents who are on haemodialysis and have itching related to long term kidney disease

Secondary aim: To measure the amount of difelikefalin that enters the blood in adolescents who are on haemodialysis and have itching related to long term kidney disease

Study Design At least 18 adolescents, aged 12 to 17 years, who are on haemodialysis and have itching related to long term kidney disease will take part in this study.

All study participants will receive difelikefalin 3 (or up to 4) times weekly for up to 12 weeks. The study duration for a participant is up to 17 to 18 weeks; during this period, participants will visit the clinic 3 times weekly (during their haemodialysis visits).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability, as assessed by incidence of AEs, of 0.5 μg/kg IV difelikefalin in adolescent participants on HD (3 times weekly) with moderate-to-severe pruritus over 12 weeks. Additionally, difelikefalin plasma concentrations (Cmax and Ctrough) after multiple administrations will be evaluated at a few selected time points and the efficacy of difelikefalin in improving itching and health-related QoL will be investigated as exploratory.

Study details include:

* The study duration for a single participant will be up to 17 to 18 weeks.
* The treatment duration for each participant will be up to 12 weeks.
* The visit frequency will be 3 times weekly (during HD visits).

Trial Population:

Participants in this study must:

* Be male or female adolescent participants ≥12 to <18 years of age at the time of informed consent/assent
* Have CKD-aP on HD (at least 3 hours in duration 3 times weekly, for at least 12 weeks prior to the informed consent procedure)
* Be able to continue HD without changing its frequency or method
* Have a mean value WI-NRS score during the run-in period of >4.0 (moderate-to-severe pruritus)

Participants in this study must not:

* Be planned to receive a kidney transplant during the study
* Have known severe hepatic impairment (e.g., Child-Pugh Class C) or concurrent hepatic cirrhosis, serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the reference upper limit of normal (ULN), significant systolic or diastolic heart failure, or concurrent malignancy (except excised basal cell or squamous cell carcinoma of the skin, or carcinoma in situ that has been excised or resected completely)

Number of Participants:

At least 18 participants evaluable for the primary safety endpoint will be enrolled in the study. Note: Enrolled means participants, or their legally acceptable representatives, agreement to participate in a clinical study following completion of the informed consent process and screening. A participant will only be considered enrolled if the informed consent/assent is not withdrawn prior to participating in any study activity after screening including the run-in period.

Study Arms and Duration:

* This is a single-arm, open-label study. All participants will receive IV difelikefalin at a dose of 0.5 μg/kg of dry body weight after each HD treatment 3 times weekly for 12 weeks.
* The study includes a screening period of up to 4 weeks (including a 7-day run-in period during the week prior to enrolment), a study treatment period of 12 weeks, and a follow-up period of 7 (up to 10) days.
* If for any reason difelikefalin is interrupted for more than 1 week, the participant should be withdrawn from the study intervention.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participant must be ≥12 to <18 years of age at the time of informed consent.
* 2. Participants with CKD on HD 3 times weekly for at least 12 weeks prior to the informed consent procedure who can continue HD without changing its frequency or method.
* 3. Participants whose WI-NRS score in the 7-day run-in period (meets both of the below:
* a) WI-NRS scores have been recorded for at least 4 days through a 7-day run-in period.
* b) The mean value of the recorded WI-NRS scores is >4.0
* 4. Over the last 3 months prior to screening, the participant has had at least 1 of the following:
* a) At least 2 single-pool Kt/V measurements ≥1.2 on different dialysis days
* b) At least 2 urea reduction ratio measurements ≥65% on different dialysis days
* c) 1 single-pool Kt/V measurement ≥1.2 and 1 urea reduction ratio measurement ≥65% on different dialysis day
* 5. Prescription dry body weight ≥20 kg
* 6. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* 7. Participant and/or legal guardian (as required) is capable of providing the appropriate signed informed consent and where appropriate, assent.

Exclusion Criteria:

* 1. Known to be non-compliant with HD treatments and deemed unlikely by the Investigator to complete the study
* 2. Planned to receive a kidney transplant during the study. Note: being listed on a kidney transplant list is not an exclusion criterion.
* 3. Participants with itching caused by conditions other than chronic renal failure or complications of chronic renal failure, which could in the opinion of the Investigator affect the efficacy evaluation (e.g., atopic dermatitis, chronic urticaria).
* 4. Participants with localised itch restricted to the palms of the hands.
* 5. Participants with pruritus only during the dialysis session (by participant report).
* 6. Participants with known concurrent hepatic cirrhosis or severe hepatic impairment (e.g., Child-Pugh Class C).
* 7. Significant systolic or diastolic heart failure (e.g., New York Heart Association Class IV congestive heart failure).
* 8. Participants with concurrent malignancy except excised basal cell or squamous cell carcinoma of the skin, or carcinoma in situ that has been excised or resected completely.
* 9. Severe mental illness or cognitive impairment (e.g., dementia) or other concurrent mental disorder that, in the opinion of the Investigator, would compromise the validity of study measurements.
* 10. Conditions associated with clinically important disruptions to the blood brain barrier (for example, primary brain malignancies, CNS metastases or other inflammatory conditions, active multiple sclerosis, advanced Alzheimer's disease) that in the Investigator's opinion may be associated with unacceptable risk for CNS effects.
* 11. Acute or unstable medical condition(s) that in the Investigator's opinion, may be associated with increased risk to the participant, or may interfere with study assessments, outcomes, or the ability to provide written informed consent or comply with study procedures.
* 12. Participant is receiving ongoing ultraviolet B treatment and anticipates receiving such treatment during the study.
* 13. New or change of treatment received for itch including antihistamines and corticosteroids (oral, IV, or topical) within 14 days prior to screening.
* 14. New or change of prescription for opioids, gabapentin, or pregabalin within 14 days prior to screening.
* 15. Participant is receiving prohibited medication (e.g., nalfurafine hydrochloride, opioid antagonists) that cannot be stopped at least 14 days before enrolment in the study.
* 16. Participant has known hypersensitivity to the study intervention or any components of the difelikefalin formulation.
* 17. Known or suspected history of alcohol, narcotic, or other drug abuse or substance dependence within 12 months prior to screening or participant with any alcoholic beverage intake of more than two units per day more than once per week.
* 18. Participation in any other investigational device or drug study <30 days prior to screening, or current treatment with other investigational agent(s).
* 19. Serum ALT, AST greater than 3× the reference ULN.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 18 weeks
  To evaluate the safety of 0.5 μg/kg difelikefalin in HD adolescents (≥12 to <18 years) with moderate-to-severe pruritus

SECONDARY OUTCOMES:
Pre-dose difelikefalin plasma concentrations (Cpre) | 12 weeks
  To evaluate difelikefalin plasma concentrations after multiple administrations of 0.5 μg/kg difelikefalin in HD adolescents (≥12 to <18 years) with moderate-to-severe pruritus
Trough difelikefalin plasma concentrations (Ctrough) | 12 Weeks
  To evaluate difelikefalin plasma concentrations after multiple administrations of 0.5 μg/kg difelikefalin in HD adolescents (≥12 to <18 years) with moderate-to-severe pruritus
Maximum difelikefalin plasma concentrations (Cmax) | 12 Weeks
  To evaluate difelikefalin plasma concentrations after multiple administrations of 0.5 μg/kg difelikefalin in HD adolescents (≥12 to <18 years) with moderate-to-severe pruritus

CONTACTS AND LOCATIONS:
Locations (7):
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario Valle de Hebron, Barcelona
- United Kingdom (3):
  - Royal Hospital for Children Glasgow - 82600073, Glasgow
  - Manchester University NHS Foundation Trust, Glasgow
  - Alder Hey Childrens Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.